CLINICAL TRIAL: NCT04347967
Title: The Safety and Tolerability After Intravenous Infusion of UMC119-06 in Subjects With Acute Respiratory Distress Syndrome (ARDS).
Brief Title: Mesenchymal Stem Cells for The Treatment of Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meridigen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMC119-06-ARDS-01
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UMC119-06 (Experimental): Human Umbilical Cord Derived-Mesenchymal Stem Cells, Single treatment by intravenous infusion.
  Interventions: Biological: UMC119-06

INTERVENTIONS:
Biological: UMC119-06 — Cohort 1: Low does of UMC119-06；Cohort 2: Medium does of UMC119- 06；Cohort 3: High does of UMC119-06

SUMMARY:
The clinical study with UMC119-06 is designed to investigate the safety in patients with moderate acute respiratory distress syndrome ("ARDS"). This will be a dose escalation, open-label, single-center study in adult with ARDS. UMC119-06 is ex vivo cultured human umbilical cord derived mensenchymal stem cells (hUC-MSCs) product which is intended for treatment of ARDS.

DETAILED DESCRIPTION:
ARDS, a noncardiogenic respiratory disease, is characterized by progressive hypoxemia and respiratory distress, associated with explosive acute inflammation and alveolar edema. ARDS occurs in all age group of patients, where mortality rates increase in advancing age.

In animal studies of ARDS, mensenchymal stem cells (MSCs) can attenuate lipopolysaccharides (LPS)-induced lung injury and pulmonary permeability edema through modulating the inflammatory. These findings show that MSCs may improve the clinical outcomes and prognosis of ARDS patient. Meridigen is developing UMC119-06, human umbilical cord-derived MSCs, for the treatment of ARDS. The purpose of this study is to assess the safety of UMC119-06 in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of age ≥ 20 years and ≤ 85 years.
* Subject has a diagnosis of moderate ARDS according to the Berlin definition of ARDS:

  1. No clinical evidence of left atrial hypertension for bilateral pulmonary infiltrates.
  2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph.
  3. Hypoxemia: PaO2/ FiO2 > 100 mmHg to ≤ 200 mmHg with PEEP ≥ 5 cm H2O.
  4. The time of onset of ARDS is when all of the specified ARDS criteria (2a-c) are met.
* Patient is intubated and mechanically ventilated.
* Subjects who had an onset of ARDS within 72 to 120 hours before start of treatment.
* Subjects with body weight between 40 to 90 kg.
* No decompensated heart failure.
* Subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided.
* Women of child-bearing potential should have a negative serum pregnancy test prior to administration of investigational product., UNLESS they meet the following criteria:

  1. Post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40 mIU/ml, OR;
  2. 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy.

Exclusion Criteria:

* Greater than 72 hours since first meeting ARDS criteria per the Berlin definition.
* No intent/unwillingness to follow lung protective ventilation strategy or fluid management protocol.
* Expected life < 3 months from other cause than the respiratory failure.
* Subject is receiving extra-corporeal membrane oxygenation, high-frequency oscillatory ventilation or any form of extra-corporeal lung support.
* Subjects with history of any type of malignancy.
* Major trauma in the prior 5 days.
* Subjects with major surgery (body organs that require anesthesia, such as tumor removal, open chest, heart surgery, abdominal surgery, intracranial surgery, or normal surgery for more than 3 hours, etc.) within previous 14 days.
* Subjects who are pregnant (or plan to become pregnant within 3 months of investigational product treatment) or lactating.
* Subjects who have a significant concomitant illness as judged by principal investigator (PI).
* Subjects who have significant abnormal laboratory tests at screening:

  1. >5 × upper limit of normal for alanine aminotransferase (ALT) or aspartate aminotransferase (AST).
  2. >3 × upper limit of normal for total bilirubin.
  3. >2 × upper limit of normal for serum creatinine.
* Subjects with known human immunodeficiency virus infection or who are immune compromised.
* Subjects who are unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation.
* Subjects with a history of severe allergic or anaphylactic reactions.
* Subjects with known allergy or hypersensitivity to any component of the formulation (normal saline and human serum albumin).
* Subjects who have participated in another clinical study of new investigational therapies or have received an investigational therapy within the 12 weeks before study drug administration.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of adverse events related to administration of UMC119-06. | 3 months from the day of administration
  Incidence of Treatment-Emergent Adverse Events (TEAEs). Incidence of withdrawals due to AEs.

SECONDARY OUTCOMES:
Changes in mortality status | 15 months from the day of administration.
  Improvement in mortality status.
Ventilator Free Days (VFD) | 28 days from the day of administration
  Improvement in clinical function as assessed by Ventilator Free Days (VFD).
Change in Oxygenation Index (OI) | 7 days or discharge from ICU after the day of administration
  Improvement in clinical function as assessed by change in Oxygenation Index (OI).
Change in Lung Injury Score (LIS) | 7 days or discharge from ICU after the day of administration
  Improvement in clinical function as assessed by change in Lung Injury Score (LIS), 0-16 points, severity increasing with higher points.
Change in positive end-expiratory pressure (PEEP) | 7 days or discharge from ICU after the day of administration
  Improvement in clinical function as assessed by change in positive end-expiratory pressure (PEEP).
Change in Lung Static Compliance | 7 days or discharge from ICU after the day of administration
  Improvement in clinical function as assessed by change in Lung Static Compliance
Change in acute physiology and chronic health evaluation score (APACHE II) | 7 days from the day of administration
  Improvement in clinical function as assessed by change in acute physiology and chronic health evaluation score (APACHE II), higher scores correspond to more severe disease and a higher risk of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare., New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No